CLINICAL TRIAL: NCT01506388
Title: Foley Catheter Plus Vaginal Isosorbide Mononitrate Versus Vaginal Misoprostol for Induction of Labour:a Randomised Controlled Trial
Brief Title: A Novel Protocol for Labour Induction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed El-khayat, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12012
Record Dates: First submitted 2012-01-04; First posted 2012-01-10 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Failed Induction of Labor
Keywords: labour induction; Foley catheter; misoprostol; isosorbide mononitrate
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- folye catheter plus vaginal IMN (Experimental): intracervical foley catheter plus vaginal IMN
  Interventions: Device: foley catheter; Drug: Vaginal IMN
- Misoprostol vaginally (Active Comparator): intravaginal misoprostol
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Device: foley catheter — foley 14 catheter intracervical plus vaginal IMN 40 mg evry 6 hours
  Arms: folye catheter plus vaginal IMN
Drug: Misoprostol — misoprostol 50 Ug , vaginally every 4-6 hours
  Other Names: misoprostol vaginally
  Arms: Misoprostol vaginally
Drug: Vaginal IMN — IMN vaginal 40 mg every 4-6 hours
  Arms: folye catheter plus vaginal IMN

SUMMARY:
The use of foley catheter was tested many times and proved to be effective for induction of labour.

DETAILED DESCRIPTION:
The investigators compare between vaginal misoprostol versus foley catheter plus vaginal isosorbide mononitrate (IMN) for induction of labour

ELIGIBILITY:
Inclusion Criteria:

* Term or post term pregnancies.
* Live,singleton fetus.
* Cephalic presentation.
* Intact membrane.
* Bishop score < 6.
* Not in labour.
* Medically indicated for labour induction.
* Primigravida or parity of 3 or less.

Exclusion Criteria:

* Previous caesarean delivery.
* Malpresentation.
* Placenta previa.
* Sever intrauterine growth restriction.
* Multiple pregnancy.
* Polyhydramnios.
* Oligohydramnios.
* Bishop score 7 or more.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
caesarean section rate | 1 year
  caesarean section

SECONDARY OUTCOMES:
time from induction to delivery | 1 year
  from the insertion of the foley catheter to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-khayat, M.D., Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Cairo University, Cairo, Cairo Governorate
  - Waleed El-khayat, Cairo, Cairo Governorate

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] El-Khayat W, Alelaiw H, El-kateb A, Elsemary A. Comparing vaginal misoprostol versus Foley catheter plus vaginal isosorbide mononitrate for labor induction. J Matern Fetal Neonatal Med. 2016;29(3):487-92. doi: 10.3109/14767058.2015.1007036. Epub 2015 Feb 19. PMID 25694257